CLINICAL TRIAL: NCT03946839
Title: Mechanism of Cognitive Impairment in ICU Sepsis/Septic Shock Survivors :a Study Using Resting-stage fMRI Technique
Brief Title: Functional Magnetic Resonance Imaging (fMRI) of Brain in ICU Survivors With Cognitive Impairment
Status: Completed | Type: Observational
Sponsor: Jian-jun Yang (Other)
Responsible Party: Sponsor-Investigator, Jian-jun Yang, Director,Department of Anesthesiology, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Other Study IDs: 20190510
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Cognitive Impairment; Functional Magnetic Resonance Imaging; Septic Shock; Inflammation
MeSH Terms: conditions — Cognitive Dysfunction; Shock, Septic; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU Survivors: sepsis/septic shock Patients with high risk of cognitive impairment who discharge from ICU
- Healthy Control: The control group have to be medically and cognitively healthy. These individuals are recruited from the community and all attempts will be made to match them on age,sex and education to individuals recruited for groups of ICU Survivors.

SUMMARY:
Long-term cognitive dysfunction greatly influences patient's quality of life after critical illness. However,its neurophysiological basis remains unknown.This is a 3 year fMRI study conducted at the Jiangyin people's Hospital. This study utilize resting-state functional magnetic resonance imaging(fMRI) to investigate the regional alterations in survivors with cognitive impairment.Further, the investigators hypothesize that these regional changes in fMRI activity are predictive of cognitive impairment.

DETAILED DESCRIPTION:
Critically ill patients who had hospitalized in ICU at least 2 days and who consented to participate will take the examination of brain fMRI,blood inflammatory markers and cognitive assessment after ICU discharge. Individuals of healthy control group are recruited from the community will be made to match them on age,sex and education to individuals recruited for groups of ICU Survivors.Those healthy people will also take the examination of brain fMRI,blood inflammatory markers and cognitive assessment.

ELIGIBILITY:
Inclusion Criteria:

ICU sepsis/septic shock Survivors

* Men and women older than 18;education years≥6(could speak, read, and write);Hospitalized in the ICU more than 2 days and already discharge from ICU;

Exclusion Criteria:

* MRI incompatibility;History of neurological disease(diagnosis of depression, schizophrenia, epilepsy, Parkinson's disease, Alzheimer's disease, demyelinating disease, cerebrovascular disease,etc);Severe brain injury;History of alcohol and drug addiction;use of psychotropic medications such as sleeping pills, selective serotonin reuptake inhibitors,etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ICU sepsis/septic shock Survivors of Jiangyin people's Hospital and healthy people from community recruitment
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Brief assessment of cognitive impairment | 1.5 h before fMRI examination
  Cognitive impairment assessed with help of MMSE(Mini-mental State Examination).The MMSE has 5 scaled scores; the scores are weighted sums of the questions in each section. The 5 sections and their range of score are listed below:Orientation 0-10;Registration 0-3;Attention and calculation 0-5;Recall 0-3;Language 0-9.Total score range from 0-30. Lower scores = more disability, higher scores = less disability.
Resting-state functional magnetic resonance imaging results | Up to 1 month after ICU discharge(It was judged by the doctor in charge according to the patient's recovery)
  3D T1-weighted magnetization parameters: TR/TE/flip angle = 7.2 ms/min full/8; FOV = 256 mm; 312 slices; slice thickness = 1 mm.
  For the BOLD sequence, a series of 35 interleaved transversal slices were acquired for full-brain coverage with a gradient-echo based, echo planar imaging (EPI) sequence with the following parameters: TR/TE/ flip angle = 2000 ms/30 ms/90; FOV = 224 mm; slice thickness = 4.0 mm.
Blood inflammatory markers | 2h before taking fMRI examination
  2-4 ml of blood was drawn for blood inflammatory markers(IL-1β,IL-2R,IL-6,IL-8,TNF-α) detection.

SECONDARY OUTCOMES:
Blood markers | the same day with fMRI examination（2h before taking fMRI examination）
  2-4 ml of blood was drawn for blood markers(NSE) detection.
Assessment of cognitive impairment | 1.5h before taking fMRI examination
  Cognitive impairment assessed with help of MoCA(Montreal Cognitive Assessment).Total score range from 0-30. Lower scores = more disability, higher scores = less disability.
Specific assessment of cognitive impairment 1 | 1.5h before taking fMRI examination
  Cognitive impairment assessed with help of DS(digit span test),including DST-F(Forward digit span test) and DST-B(backward digit span test).Total score range from 5-20. Lower scores = more disability, higher scores = less disability.
Specific assessment of cognitive impairment 2 | 1.5h before taking fMRI examination
  Cognitive impairment assessed with help of AVLT(auditory verbal learning test),Total score range from 0-12. Lower scores = more disability, higher scores = less disability.
Specific assessment of cognitive impairment 3 | 1.5h before taking fMRI examination
  Cognitive impairment assessed with help of CFT(complex figure test),Total score range from 0-36. Lower scores = more disability, higher scores = less disability.
Specific assessment of cognitive impairment 4 | 1.5h before taking fMRI examination
  Cognitive impairment assessed with help of SDMT(symbol digit modalities test),Total score range from 0-105. Lower scores = more disability, higher scores = less disability.
Specific assessment of cognitive impairment 5 | 1.5h before taking fMRI examination
  Cognitive impairment assessed with help of VFT(verbal fluency test),The total score was the number of animals named in one minute. Lower scores = more disability, higher scores = less disability.
Specific assessment of cognitive impairment 6 | 1.5h before taking fMRI examination
  Cognitive impairment assessed with help of CDT(clock drawing test),Total score range from 0-4. Lower scores = more disability, higher scores = less disability.
Specific assessment of cognitive impairment 7 | 1.5h before taking fMRI examination
  Cognitive impairment assessed with help of TMT-A(trail making test part A) and TMT-B(trail making test part B), the test outcome was the time to complete the test(seconds). Longer time = more disability, Shorter time = less disability.
Assessment of Depression | 1.5h before taking fMRI examination
  SDS(self-rating depression scale) was used to assess the depression status of the participants in the past week.The SDS has 20 questions; each question was scored on a scale of 1-4;total score range from 20-80;the standard score(total score multiplied by 1.25):less than 53 was normal group,53-62 was mild depression, 63-72 was moderate depression, more than 72 was severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Mu huo Ji, PhD, Principal Investigator — Zhongda Hospital
Locations (1):
- Jiangyin People's Hospital, Jiangyin, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
Most participants were reluctant to share their personal information with researchers outside this study.